CLINICAL TRIAL: NCT05662644
Title: Minimally Invasive Surgery for Esophageal Cancer: Feasibility and Outcome
Brief Title: Assessment of Minimally Invasive Surgery for Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Abd Elraheem Mohamed Kenawy, teaching assistant, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-11-10
Record Dates: First submitted 2022-12-05; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Esophageal Cancer
Keywords: Minimally invasive; Esophageal Cancer; feasibility; outcome
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Intervention Model Description: All patients with esophageal cancer who are considered candidates for esophagectomy present to NCI in the period starting fromDecember 2022
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feasibility of Esophagectomy Esophageal Cancer (Active Comparator): Minimally Invasive Surgery for Esophageal Cancer: feasibility
  Interventions: Procedure: Minimally Invasive Surgery for Esophageal Cancer
- Outcome of Esophagectomy Esophageal Cancer (Active Comparator): Minimally Invasive Surgery for Esophageal Cancer: outcome
  Interventions: Procedure: Minimally Invasive Surgery for Esophageal Cancer

INTERVENTIONS:
Procedure: Minimally Invasive Surgery for Esophageal Cancer — Assessment of minimally Invasive Surgery for Esophageal Cancer

SUMMARY:
Evaluate the feasibility and outcome of minimally invasive management of esophageal cancer regarding

1. Surgical technique:

   A totally minimally invasive technique (combined thoracoscopic and laparoscopic approaches) for esophagectomy will be used in this study. Also, a hybrid technique (thoracoscopic approach with laparotomy or laparoscopic approach with thoracotomy) will be included.
2. Histopathology

   * Assessment of surgical margins
   * Assessment of the number of lymph nodes
3. Peri-operative outcome including

   * Operative time
   * Conversion to open
   * Blood loss
   * Hospital stays
4. Evaluation of recurrence, disease-free survival and overall survival rates: according to The Kaplan-Meier estimator
5. Morbidity and mortality.

DETAILED DESCRIPTION:
Introduction

Esophageal cancer is the seventh most common cause of cancer-related death worldwide. The overall five-year survival is below 20%.

It is characterized by its high mortality rate, poor prognosis at time of diagnosis and variability based on geographic location. Now , the prevalence of esophageal cancer is in transition .

The Arabic world has very low incidences of Esophageal cancer in general. In Egypt, it represents 1.7% of all cancers.

Esophagectomy followed by reconstruction surgery has been the most reliable modality for treatment in patients without evidence of disease spread.

Different surgical approaches, such as the Sweet esophagectomy, Ivor Lewis esophagectomy, McKeown esophagectomy, and transhiatal esophagectomy, have been used clinically based on specific locations in the esophageal cancer.

For cancer of the middle or lower segment of the thoracic esophagus, the Ivor Lewis esophagectomy and the Sweet esophagectomy through the left thoracic approach are the mainstream standard surgical approaches.

Conventional surgical treatment involves open esophagectomy (OE) using transthoracic or transhiatal approaches which are associated with high mortality and morbidity especially respiratory complications (RCs) that are common with open esophagectomy and can increase the risk of death by up to 20%.

Traditionally, an esophagectomy was performed through a right thoracotomy and laparotomy. However, these patients are at a high risk for developing postoperative pulmonary complications. In order to decrease postoperative morbidity, minimally invasive surgical techniques were introduced in the treatment of esophageal cancer.

The first thoracoscopic esophageal mobilizations for esophagectomy were performed in the early 1990s by A. Cuschieri.

Then, DePaula and colleagues and Swanström and Hansen separately published the first totally minimally invasive transhiatal esophagectomies in 1995 and 1997, respectively. Subsequently, many centers began to adapt their preferred technique to minimally invasive approaches and gained significant experience in laparoscopic and thoracoscopic approaches to esophagectomy.

Luketich et al. first identified the combined thoracoscopic esophageal mobilization followed by the laparoscopic fashioning of the gastric conduit and the development of an esophagogastric anastomosis in the cervical region.

In recent decades, minimally invasive esophagectomy (MIE) has become an alternative to open esophagectomy. minimally invasive esophagectomy (MIE) involves several techniques including total MIE (tMIE), hybrid minimally invasive esophagectomy (hMIE), and robotic surgery .

The procedure consists presently of three main techniques: combined thoracoscopic and laparoscopic approach (Ivor Lewis); thoracoscopic, laparoscopic, and cervical approach (three-hole); or laparoscopic and cervical approach only (transhiatal).

Luketich et al. subsequently published their approach to minimally invasive Ivor Lewis esophagectomy and intrathoracic anastomosis and concluded that this type of treatment is feasible.

MI McKeown esophagectomy procedure consists of thoracoscopic esophagectomy, laparoscopic gastric mobilization, and cervical anastomosis between the esophageal stump and gastric stump. With the improvement of techniques and equipment, McKeown MIE has received increased attention.

Objectives:

Evaluate the feasibility and outcome of minimally invasive management of esophageal cancer regarding

1. Surgical technique:

   A totally minimally invasive technique (combined thoracoscopic and laparoscopic approaches) for esophagectomy will be used in this study. Also, a hybrid technique (thoracoscopic approach with laparotomy or laparoscopic approach with thoracotomy) will be included.
2. Histopathology

   * Assessment of surgical margins
   * Assessment of the number of lymph nodes
3. Peri-operative outcome including

   * Operative time
   * Conversion to open
   * Blood loss
   * Hospital stays
4. Evaluation of recurrence, disease-free survival and overall survival rates: according to The Kaplan-Meier estimator
5. Morbidity and mortality.

Aim of the work This study aims to evaluate the feasibility and outcome of minimally invasive management of esophageal cancer.

Study Design:

This study is going to be a prospective study where patients presenting with esophageal cancer who are considered candidates for surgery will undergo minimally invasive surgery. Each patient will be assessed in the pre, intra, and short postoperative period.

Methodology:

1. Population of study & disease Condition patients with esophageal cancer.
2. Background and Demographic characteristics Any patient with esophageal cancer is considered a candidate for a minimally invasive esophagectomy procedure.
3. Inclusion criteria:

   * Any age.
   * Any sex.
   * Diagnostic operable esophageal cancer.
4. Exclusion criteria:

   * Metastatic patients.
   * Locally advanced cases.
   * Patients with comorbidities who are unfit for major surgical procedures.
   * Patients with contraindications for laparoscopy or thoracoscopy.
5. Interventions:

   Patients with esophageal cancer who are considered candidates for surgery will be subjected to minimally invasive procedures through a combined laparoscopic and thoracoscopic approach with D2 dissection and mediastinal dissection.
6. Possible Risk:

   The main risks are the same as Open esophagectomy Procedures as surgical site complications, pulmonary complications, bleeding, Leakage, mediastinitis, fluid collection, and stenosis.

   Also, there is a risk of conversion from minimally invasive to open technique.
7. Primary outcome parameters:

   The primary outcome will be the assessment of operative time, hospital stay, intraoperative and early postoperative complications, and the assessment of pathology regarding surgical margins and the retrieved lymph nodes.
8. Secondary outcome parameters:

   The secondary outcome will be the incidence of late complications such as anastomotic stenosis and reflux symptoms and also the incidence of locoregional recurrence.
9. Sample size (number of participants included) All patients with esophageal cancer who are considered candidates for esophagectomy present to NCI in the period of 2 years starting November 2022 till October 2024.
10. Statistical analysis:

    Data will be collected in preformed data collection before being entered in the spreadsheet. Statistical analysis will be performed using the statistical package for social science (SPSS). Continuous variables will be expressed as mean and standard deviation (normally distributed data) or median and range (not normally distributed data) while categorical data expressed as numbers and percentages.

    Chi-square test will be used to compare the nominal data while continuous data will be compared by the student t-test (normally distributed data) and Mann-Whitney test (not normally distributed data).
11. Source of funding:

Self-funding.

ELIGIBILITY:
Inclusion Criteria:

* Any age.
* Any sex.
* Diagnostic operable esophageal cancer.

Exclusion Criteria:

* Metastatic patients.
* Locally advanced cases.
* Patients with comorbidities who are unfit for major surgical procedures.
* Patients with contraindications for laparoscopy or thoracoscopy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Duration of Operatiion | 1 day postoperative
  minutes
Duration of hospital stay | 2 weeks postoperative
  Days
Type of Surgical technique | 1 day postoperative
  Thoracoscopic, laparoscopic or combined
Status of surgical margins | 2 weeks postoperative
  Free or not
Number of lymph nodes | 2 weeks postoperative
  numbers
occurence of Conversion to open | 1 day postoperative
  yes or no
Amount of Blood loss | 1 day postoperative
  Milliliters
Incidence of recurrence | 6 months postoperative
  yes or no
Occurrence of intraoperative vascular injury | 1 day postoperative
  yes or no
Occurence of anastomotic leakage | 4 weeks postoperative
  yes or no
Administration of neoadjuvant therapy | 2 weeks preoperative
  yes or no
Level of preoperative Haemoglobin | 1 week preoperative
  g/dl
Level of postoperative Haemoglobin | 1 week postoperative
  g/dl
Level of CEA preoperative | 2 weeks preoperative
  ng/ml
Level of CEApostoperative | 4 weeks postoperative
  ng/ml
Occurence lung injury | 1 day postoperative
  yes or no
site of pathology | 1 day preoperative
  upper / middle or lower esophageal
type of anastomosis | 1 day postoperative
  stapler or hand sewing
Nature of gross picture of specimen | 2 weeks postoperative
  mass / ulcer

SECONDARY OUTCOMES:
Occurence of mortality | 6 weeks postoperative
  yes or no
Occurence of anastomotic stenosis | 6 weeks postoperative
  yes or no
Occurence of ostoperative reflux | 6 weeks postoperative
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Kenawy, MD, Principal Investigator — Sohag University; Alaa-Eldin H Mohamed, professor, Study Chair — Sohag University; Alaa A Redwan, professor, Study Director — Sohag University; Haitham F Othman, MD, Study Director — National Cancer Institute (NCI)
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided